CLINICAL TRIAL: NCT06481891
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study to Evaluate the Efficacy and Safety of SOtaglifloziN in symptomATic Obstructive And Non-obstructive Hypertrophic CardioMyopathy (SONATA-HCM)
Brief Title: A Study to Evaluate the Efficacy and Safety of Sotagliflozin in Symptomatic Obstructive and Non-obstructive Hypertrophic Cardiomyopathy
Acronym: SONATA-HCM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LX4211.1-314-HCM
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Obstructive Cardiomyopathy, Hypertrophic; Non-obstructive Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sotagliflozin (Experimental): Following an up to 3-week screening period, sotagliflozin 400 milligrams (mg) tablets will be administered as two 200 mg tablets, once daily, before the first meal of the day in the double-blind treatment period for up to 26 weeks.
  Interventions: Drug: Sotagliflozin
- Placebo (Placebo Comparator): Following an up to 3-week screening period, sotagliflozin-matching placebo 400 mg tablets will be administered as two 200 mg tablets, once daily, before the first meal of the day in the double-blind treatment period for up to 26 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sotagliflozin — Sotagliflozin will be administered as a tablet(s), orally once daily.
  Other Names: SAR439954/LX4211
  Arms: Sotagliflozin
Drug: Placebo — Placebo will be administered as a tablet(s) (identical to the sotagliflozin tablet in appearance), orally once daily.
  Other Names: SAR439954/LX4211
  Arms: Placebo

SUMMARY:
The main purpose of the study is to determine the changes in symptoms and functional limitations in participants with symptomatic hypertrophic cardiomyopathy (HCM) treated with sotagliflozin as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* KCCQ CSS < 85.
* NYHA functional class II or III
* A diagnosis of HCM consistent with the current American College of Cardiology Foundation/American Heart Association and European Society of Cardiology guideline definition: unexplained left ventricular (LV) hypertrophy with nondilated ventricular chambers in the absence of other cardiac (eg, hypertension, aortic stenosis) or systemic disease with maximal LV wall thickness ≥ 15 millimeters (mm), or ≥ 13 mm with positive family history of HCM.
* For obstructive hypertrophic cardiomyopathy (oHCM), left ventricular outflow tract (LVOT) peak gradient ≥ 30 millimetre of mercury (mm Hg) during screening as assessed by echocardiography at rest or during a valsalva maneuver.
* For nonobstructive hypertrophic cardiomyopathy (nHCM), LVOT peak gradient < 30 mm Hg during screening as assessed by echocardiography at rest and < 30 mm Hg during a valsalva maneuver.
* Screening left ventricular ejection fraction (LVEF) ≥ 50%, except for those on a cardiac myosin inhibitor (screening LVEF ≥ 55%).
* For participants on a cardiac myosin inhibitor, the dose must be stable at least 3 months prior to screening. Participants on cardiac myosin inhibitor should not be scheduled for up-titration during the trial.
* Stable doses of background therapy (ie, β-blockers, calcium channel blockers, angiotensin-converting enzyme (ACE) inhibitors, angiotensin receptor blockers, diuretics) for at least 1 month prior to screening.

Exclusion Criteria:

* Received therapy with a sodium glucose co-transporter 2 (SGLT2) inhibitor within the past 8 weeks prior to screening.
* Previous intolerance to an SGLT2 inhibitor.
* Any previous treatment with sotagliflozin.
* Current use of thiazolidinediones or digoxin.
* Current/planned participation in another interventional clinical trial or prior participation in any interventional trial with an investigational agent within 45 days of screening.
* Known infiltrative or storage disorder causing cardiac hypertrophy that mimics HCM such as Fabry disease, amyloidosis, or Noonan syndrome with LV hypertrophy.
* History of unexplained syncope within 6 months prior to screening.
* History of sustained ventricular tachyarrhythmia (> 30 seconds) or appropriate implantable cardioverter defibrillator (ICD) discharge within 6 months prior to screening.
* Has paroxysmal, persistent, or permanent atrial fibrillation not on anticoagulation for at least 4 weeks prior to screening and/or not adequately rate controlled within 3 months of screening.
* Septal reduction therapy planned during the study period. For participants who had septal reduction therapy, the procedure should have been completed more than 3 months prior to screening.
* Cardiac surgery (eg, coronary artery bypass graft, valvular repair/replacement), percutaneous coronary intervention, or implantation of cardiac device (pacemaker or implantable cardioverter defibrillator) within 3 months prior to screening or planned during the study period.
* Presence of a cardiac resynchronization therapy device.
* Acute coronary syndrome within 2 months prior to screening.
* History of stroke or myocardial infarction within 6 months prior to screening.
* Hospitalization for heart failure or arrhythmia within 4 weeks prior to screening.
* Has known moderate or severe (as per investigator's judgment) aortic valve stenosis at screening.
* Current angina or clinically significant ischemia due to unstable epicardial coronary disease, as per investigator judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to Week 26 in Kansas City Cardiomyopathy Questionnaire Clinical Summary Score (KCCQ CSS) | Baseline to Week 26
  KCCQ is a 23-item, self-administered questionnaire that measure the participant's perception of their health status, including their heart failure (HF) symptoms, impact on physical and social function and how their HF impacts the quality of life. KCCQ quantifies 7 domains: physical limitations (6 items), symptom stability (1 item), symptom frequency (4 items), symptom burden (3 items), self-efficacy (2 items), quality of life (3 items) and social limitations (4 items). Scores are generated for each domain and scaled from 0 to 100, with 0 denoting the worst and 100 the best possible status. Higher scores reflect better health status.

SECONDARY OUTCOMES:
Percentage of Participants at Week 26 with a New York Heart Association (NYHA) Functional Class Improvement ≥ 1 Category | Week 26
  NYHA functional class is a clinician-reported assessment of participants' health status on a 4-point scale, where Class I represents no limitations in normal activity; Class II indicates slight limitation of physical activity; Class III indicates marked limitation in physical activity; and Class IV indicates that participants have symptoms with any physical activity or at rest. Percentage of participants with NYHA functional class improvement ≥1 will be reported.
Change from Baseline to Week 26 in KCCQ Total Symptom Score (TSS). | Baseline to Week 26
  KCCQ is a 23-item, self-administered questionnaire that measure the participant's perception of their health status, including their HF symptoms, impact on physical and social function and how their HF impacts the quality of life. KCCQ quantifies 7 domains: physical limitations (6 items), symptom stability (1 item), symptom frequency (4 items), symptom burden (3 items), self-efficacy (2 items), quality of life (3 items) and social limitations (4 items). Scores are generated for each domain and scaled from 0 to 100, with 0 denoting the worst and 100 the best possible status. Higher scores reflect better health status.

CONTACTS AND LOCATIONS:
Locations (103):
- United States (30):
  - Lexicon Investigational Site (4037), Scottsdale, Arizona
  - Lexicon Investigational Site (4012), Los Angeles, California
  - Lexicon Investigational Site (4035), Pomona, California
  - Lexicon Investigational Site (4044), San Francisco, California
  - Lexicon Investigational Site (4034), Orlando, Florida
  - Lexicon Investigational Site (4018), Atlanta, Georgia
  - Lexicon Investigational Site (4033), Evanston, Illinois
  - Lexicon Investigational Site (4036), Merrillville, Indiana
  - Lexicon Investigational Site (4021), Baltimore, Maryland
  - Lexicon Investigational Site (4016), Boston, Massachusetts
  - Lexicon Investigational Site (4042), Boston, Massachusetts
  - Lexicon Investigational Site (4028), Ann Arbor, Michigan
  - Lexicon Investigational Site (4038), Grand Rapids, Michigan
  - Lexicon Investigational Site (4027), Rochester, Minnesota
  - Lexicon Investigational Site (4013), St Louis, Missouri
  - Lexicon Investigational Site (4029), Morristown, New Jersey
  - Lexicon Investigational Site (4039), Manhasset, New York
  - Lexicon Investigational Site (4043), New York, New York
  - Lexicon Investigational Site (4026), Morrisville, North Carolina
  - Lexicon Investigational Site (4031), Cincinnati, Ohio
  - Lexicon Investigational Site (4017), Cleveland, Ohio
  - Lexicon Investigational Site (4024), Tulsa, Oklahoma
  - Lexicon Investigational Site (4015), Portland, Oregon
  - Lexicon Investigational Site (4011), Philadelphia, Pennsylvania
  - Lexicon Investigational Site (4019), Germantown, Tennessee
  - Lexicon Investigational Stie (4014), Houston, Texas
  - Lexicon Investigational Site (4032), Charlottesville, Virginia
  - Lexicon Investigational Site (4010), Seattle, Washington
  - Lexicon Investigational Site (4022), Marshfield, Wisconsin
  - Lexicon Investigational Site (4040), Milwaukee, Wisconsin
- Argentina (7):
  - Lexicon Investigational Site (5016), Santa Rosa, La Pampa Province
  - Lexicon Investigational Site (5012), Rosario, Santa Fe Province
  - Lexicon Investigational Site (5015), Corrientes
  - Lexicon Investigational Site (5010), Córdoba
  - Lexicon Investigational Site (5013), Córdoba
  - Lexicon Investigational Site (5011), Salta
  - Lexicon Investigational Site (5014), Santa Fe
- Lexicon Investigational Site (1012), Genk, Belgium
- Brazil (4):
  - Lexicon Investigational Site (5114), Salvador, Estado de Bahia
  - Lexicon Investigational Site (5110), Campinas, São Paulo
  - Lexicon Investigational Site (5112), Recife
  - Lexicon Investigational Site (5115), São Paulo
- Bulgaria (2):
  - Lexicon Investigational Site (1112), Rousse
  - Lexicon Investigational Site (1111), Sofia
- Croatia (4):
  - Lexicon Investigational Site (1215), Krapinske Toplice
  - Lexicon Investigational Site (1212), Opatija
  - Lexicon Investigational Site (1210), Rijeka
  - Lexicon Investigational Site (1213), Zagreb
- Czechia (3):
  - Lexicon Investigational Site (1311), Brno
  - Lexicon Investigational Site (1310), Prague
  - Lexicon Investigational Site (1312), Ústí nad Labem
- France (6):
  - Lexicon Investigational Site (1514), Chambray-lès-Tours
  - Lexicon Investigational Site (1511), Marseille
  - Lexicon Investigational Site (1513), Paris
  - Lexicon Investigational Site (1510), Poitiers
  - Lexicon Investigational Site (1512), Rennes
  - Lexicon Investigational Site (1515), Toulouse
- Georgia (4):
  - Lexicon Investigational Site (1611), Tbilisi
  - Lexicon Investigational Site (1610), Tbilisi
  - Lexicon Investigational Site (1612), Tbilisi
  - Lexicon Investigational Site (1613), Tbilisi
- Germany (4):
  - Lexicon Investigational Site (2813), Berlin
  - Lexicon Investigational Site (2812), Hamburg
  - Lexicon Investigational Site (2811), Leipzig
  - Lexicon Investigational Site (2810), München
- Hungary (4):
  - Lexicon Investigational Site (1710), Budapest
  - Lexicon Investigational Site (1711), Pécs
  - Lexicon Investigational Site (1712), Szeged
  - Lexicon Investigational Site (1713), Zalaegerszeg
- Israel (8):
  - Lexicon Investigational Site (7017), Be’er Ya‘aqov
  - Lexicon Investigational Site (7013), Haifa
  - Lexicon Investigational Site (7014), Haifa
  - Lexicon Investigational Site (7015), Holon
  - Lexicon Investigational Site (7011), Jerusalem
  - Lexicon Investigational Site (7016), Petah Tikva
  - Lexicon Investigational Site (7012), Ramat Gan
  - Lexicon Investigational Site (7019), Tel Aviv
- Italy (3):
  - Lexicon Investigational Site (1814), Arezzo
  - Lexicon Investigational Site (1811), Brescia
  - Lexicon Investigational Site (1813), Napoli
- Poland (3):
  - Lexicon Investigational Site (2113), Lodz
  - Lexicon Investigational Site (2115), Oświęcim
  - Lexicon Investigational Site (2110), Wroclaw
- Portugal (6):
  - Lexicon Investigational Site (2210), Braga
  - Lexicon Investigational Site (2213), Faro
  - Lexicon Investigational Site (2211), Lisbon
  - Lexicon Investigational Site (2215), Lisbon
  - Lexicon Investigational Site (2216), Lisbon
  - Lexicon Investigational Site (2217), Porto
- Romania (4):
  - Lexicon Investigational Site (2910), Baloteşti
  - Lexicon Investigational Site (2913), Suceava
  - Lexicon Investigational Site (2911), Târgu Mureş
  - Lexicon Investigational Site (2912), Târgu Mureş
- Serbia (5):
  - Lexicon Investigational Site (2312), Belgrade
  - Lexicon Investigational Site (2314), Belgrade
  - Lexicon Investigational Site (2311), Belgrade
  - Lexicon Investigational Site (2313), Belgrade
  - Lexicon Investigational Site (2310), Niš
- Lexicon Investigational Site (2510), Stockholm, Sweden
- United Kingdom (4):
  - Lexicon Investigational Site (2712), Glasgow
  - Lexicon Investigational Site (2713), Leicester
  - Lexicon Investigational Site (2710), Liverpool
  - Lexicon Investigational Site (2711), London

IPD SHARING:
Plan to Share IPD: No